CLINICAL TRIAL: NCT03224754
Title: Understanding Management and Clinical Follow-up of Atypia of Undetermined Significance / Follicular Lesion of Undetermined Significance Category in Thyroid Fine Needle Aspiration: A 6 Year-retrospective Study in a Tertiary Care Center.
Brief Title: Atypia of Undetermined Significance (AUS) / Follicular Lesion of Undetermined Significance (FLUS)
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Maria F. Gonzalez, Assisstant Professor of the department of Pathology, University of Mississippi Medical Center
Other Study IDs: 2017-0075
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Diagnoses Disease
Keywords: Atypia, thyroid, malignancy
MeSH Terms: conditions — Thyroid Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Determination of risk of malignancy of these thyroid lesions — This is a retrospective study that will help us to find out the rate of AUS/ FLUS in our population of Mississippi and the percentage of malignancies in these cases.The specimens will be searched through the University of Mississippi Medical Center's Pathology Laboratory Information system (Copath), from April 2010 to December 2016. The retrospective cases will be retrieved using natural language search. The total number of thyroid FNA will be retrieved and the percentage of cases with AUS/ FLUS will be calculated. Followup of these cases will be done looking for additional fine needle aspirations of the thyroid or thyroidectomy specimens. Cases with diagnosis of AUS/ FLUS will have correlation with the diagnosis on the thyroidectomy specimens if available in our system.

SUMMARY:
According to the guidelines for reporting thyroid fine needle aspirations known as The Bethesda System, the category of atypical cells known as AUS/ FLUS category has an estimated rate of 5 to 15% for malignancy. This study aims to determine the rate of malignancy of this category in our institution and to evaluate the clinical outcome of the participants.

DETAILED DESCRIPTION:
This is a retrospective study that will help us to find out the rate of AUS/ FLUS in our population of Mississippi and the percentage of malignancies in these cases.The specimens will be searched through the University of Mississippi Medical Center's Pathology Laboratory Information system (Copath), from April 2010 to December 2016. The retrospective cases will be retrieved using natural language search. The total number of thyroid FNA will be retrieved and the percentage of cases with AUS/ FLUS will be calculated. Followup of these cases will be done looking for additional fine needle aspirations of the thyroid or thyroidectomy specimens. Cases with diagnosis of AUS/ FLUS will have correlation with the diagnosis on the thyroidectomy specimens if available in our system.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid fine needle aspirations interpreted as AUS/ FLUS at University of Mississippi Medical Center from April 2010 to December 2016.

Exclusion Criteria:

* Fine needle aspirations of thyroid with diagnosis of unsatisfactory, benign, suspicious for follicular neoplasm/ Follicular neoplasm, suspicious for malignancy and malignant.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient that has a diagnosis of atypia of undetermined significance/ follicular lesion of undetermined significance after thyroid fine needle aspiration regardless the age, sex or any other condition.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Number of malignant cases in a subsequent thyroidectomy after a diagnosis of AUS/ FLUS | From April 1st/ 2010 to December 31st 2016
  All the cytology cases with a diagnosis of AUS/FLUS on fine needle aspiration from April 1st 2010 to December 31st 2016 will be retrieved using the University Medical Center's pathology information system (Copath). Follow-up of these cases will be done looking for percentage of malignancy in these cases.

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Gonzalez, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jo VY, Stelow EB, Dustin SM, Hanley KZ. Malignancy risk for fine-needle aspiration of thyroid lesions according to the Bethesda System for Reporting Thyroid Cytopathology. Am J Clin Pathol. 2010 Sep;134(3):450-6. doi: 10.1309/AJCP5N4MTHPAFXFB. PMID 20716802
- [Result] Baloch ZW, Cibas ES, Clark DP, Layfield LJ, Ljung BM, Pitman MB, Abati A. The National Cancer Institute Thyroid fine needle aspiration state of the science conference: a summation. Cytojournal. 2008 Apr 7;5:6. doi: 10.1186/1742-6413-5-6. No abstract available. PMID 18394201
- [Result] Cibas ES, Ali SZ. The Bethesda System for Reporting Thyroid Cytopathology. Thyroid. 2009 Nov;19(11):1159-65. doi: 10.1089/thy.2009.0274. PMID 19888858
- [Result] Marchevsky AM, Walts AE, Bose S, Gupta R, Fan X, Frishberg D, Scharre K, Zhai J. Evidence-based evaluation of the risks of malignancy predicted by thyroid fine-needle aspiration biopsies. Diagn Cytopathol. 2010 Apr;38(4):252-9. doi: 10.1002/dc.21185. PMID 19813257
- [Result] Renshaw A. An estimate of risk of malignancy for a benign diagnosis in thyroid fine-needle aspirates. Cancer Cytopathol. 2010 Aug 25;118(4):190-5. doi: 10.1002/cncy.20092. PMID 20586117
- [Result] Ho AS, Sarti EE, Jain KS, Wang H, Nixon IJ, Shaha AR, Shah JP, Kraus DH, Ghossein R, Fish SA, Wong RJ, Lin O, Morris LG. Malignancy rate in thyroid nodules classified as Bethesda category III (AUS/FLUS). Thyroid. 2014 May;24(5):832-9. doi: 10.1089/thy.2013.0317. Epub 2014 Mar 10. PMID 24341462
- [Result] Kim TH, Jeong DJ, Hahn SY, Shin JH, Oh YL, Ki CS, Kim JW, Jang JY, Cho YY, Chung JH, Kim SW. Triage of patients with AUS/FLUS on thyroid cytopathology: effectiveness of the multimodal diagnostic techniques. Cancer Med. 2016 May;5(5):769-77. doi: 10.1002/cam4.636. Epub 2016 Jan 18. PMID 26775803
- [Result] Singh RS, Wang HH. Eliminating the "Atypia of Undetermined Significance/Follicular Lesion of Undetermined Significance" category from the Bethesda System for Reporting Thyroid Cytopathology. Am J Clin Pathol. 2011 Dec;136(6):896-902. doi: 10.1309/AJCPIX52MBOKTICP. PMID 22095375
- [Result] Yoo MR, Gweon HM, Park AY, Cho KE, Kim JA, Youk JH, Son EJ. Repeat Diagnoses of Bethesda Category III Thyroid Nodules: What To Do Next? PLoS One. 2015 Jun 26;10(6):e0130138. doi: 10.1371/journal.pone.0130138. eCollection 2015. PMID 26115096